CLINICAL TRIAL: NCT05375214
Title: A Pilot Study of iTBS in Bipolar I Depression
Brief Title: iTBS in Bipolar I Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Baszucki Brain Research Fund (Other); Magnus Medical (Industry); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00327675
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Bipolar Depression; Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Other): Open label study, all participants will receive novel iTBS
  Interventions: Device: Magnus Transcranial Magnetic Neuromodulation System (MNS) with SAINT®(Stanford Accelerated Intelligent Neuromodulation Therapy)

INTERVENTIONS:
Device: Magnus Transcranial Magnetic Neuromodulation System (MNS) with SAINT®(Stanford Accelerated Intelligent Neuromodulation Therapy) — Novel intermittent theta burst stimulation protocol with individualized targets in the brain for stimulation using structural and functional MRI inputs

SUMMARY:
A multisite, open label pilot study to investigate the efficacy and safety of a novel accelerated intermittent theta-burst stimulation (iTBS) protocol while assessing for changes in neuroimaging biomarkers associated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. 22-65 years of age
2. Bipolar I disorder diagnosis as defined by The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
3. Currently experiencing a Major Depressive Episode with Montgomery-Asberg Depression Rating Scale (MADRS) >/= 20 at screening [Day -5/-14] and baseline [Day 0]
4. On a stable and adequate dose of an anti-manic agent (Lithium with a level of at least 0.6, Depakote with a level of at least 50, or a therapeutic dose of carbamazepine, oxcarbazepine, or a neuroleptic for treatment of mania per clinician judgment) without dose changes for at least 6 weeks prior to the active study time period. Final assessment of appropriateness of participant's pharmacologic regimen is subject to study team clinician judgment.
5. Having failed a therapeutic trial of a first line bipolar depression antidepressant (as specified by the Antidepressant Treatment History Form and updated with new medications approved by the FDA for treatment of bipolar depression) in this current episode. This includes a minimum 4 week trial of one of the following medications (minimum dosage): lithium 900mg daily (or blood level >= 0.6 milliequivalent/Liter (mEq/L), carbamazepine 400mg daily (or blood level >= 0.8 mEq/L), lamotrigine 200mg daily, asenapine 20mg daily, lurasidone 20mg daily, olanzapine 10mg daily, quetiapine 300mg daily, or lumateperone 42mg daily. Final determination of a failed adequate therapeutic trial is subject to study team clinician judgement.
6. Established outpatient psychiatrist

Exclusion Criteria:

1. Female that is pregnant or breastfeeding, or of childbearing potential but not using medically acceptable birth control during study
2. Current mixed episode assessed by clinician judgment as defined by DSM-5 criteria
3. Current active substance use disorder (as defined by DSM-5) with exception of nicotine and caffeine. Participants may be subject to urine drug screen base on study team clinician judgment.
4. Participation in any clinical trial with an investigational drug or device within the last 3 month or concurrent to study participation
5. History of epilepsy, shrapnel or metal in the head or skull, cardiovascular disease/event, Obsessive Compulsive Disorder, or autism spectrum disorder
6. Clinically defined major neurological disorder; including, but not limited to, seizure disorder and history of loss of consciousness due to head injury for greater than 10 minutes, or documented evidence of brain injury
7. Active suicidal risk based on investigator's clinical judgment
8. Clinically significant unstable medical condition
9. Other condition judged by investigator that could prevent the participant from completion of the study (such as but not limited to, significant physical disability (e.g., hearing/visual deficits) to perform a neutral memory task and/or neuropsychological test battery)
10. Ferromagnetic metal implant or another contraindication to imaging in a 3 Tesla MRI
11. Electroconvulsive therapy (ECT) treatment in the past 3 months
12. Minimum of 6 months since last manic or hypomanic episode as defined by DSM-5 criteria

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zandi, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Open label study, all participants will receive novel intermittent theta-burst stimulation (iTBS) protocol, SAINT®(Stanford Accelerated Intelligent Neuromodulation Therapy)
Period: Overall Study
Arm/Group | Treatment Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Open label study, all participants will receive novel iTBS protocol, SAINT®(Stanford Accelerated Intelligent Neuromodulation Therapy)
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Montgomery-Asberg Depression Rating Scale (MADRS) Score [Mean (Standard Deviation); unit: score on a scale] — Total scores can range from 0 to 60, with higher scores indicating greater severity of depression (0-6 normal range, 7-19 mild depression, 20-34 moderate depression, >34 severe depression).
  score on a scale | 29.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a ten-item clinician rated questionnaire that helps rate the severity of depression. Total scores can range from 0 to 60, with higher scores indicating greater severity of depression (0-6 normal range, 7-19 mild depression, 20-34 moderate depression, >34 severe depression).
  MADRS score will be assessed at baseline visit and immediate follow-up visit (which occurs within 5 days after treatment end). The change in MADRS score is calculated by baseline - immediate follow-up visit score.
Time Frame: baseline and post treatment up to 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
score on a scale | 16.9 (6.7)

ADVERSE EVENTS:
Time Frame: up to 1 month
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=10)
mild headache (General disorders) | 2 — Two participants reported mild headache after treatment, one resolved spontaneously, another resolved with over the counter pain relief.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05375214/Prot_SAP_000.pdf